CLINICAL TRIAL: NCT01823536
Title: A Phase IV, Open-label, Controlled, Multi-center Study to Evaluate the 5-year Antibody Persistence Among Children Who Previously Received Novartis MenACWY Conjugate Vaccine at 2 to 10 Years of Age and to Assess the Immune Response to a Single Dose of Novartis MenACWY Conjugate Vaccine
Brief Title: Persistence of Immunogenicity of MenACWY Conjugate Vaccine 5 Years After Childhood Vaccination, and Immune Response to a Booster Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V59P20E1
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Meningococcal Disease
Keywords: Meningitis
MeSH Terms: conditions — Meningococcal Infections; Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- MenACWY-CRM (≥7-≤10 years of age) (Experimental): Subjects, who had previously received 2 injections of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine at 2-5 years of age, were administered 1 injection of the same vaccine at 7-10 years of age.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine
- MenACWY-CRM_1 (≥7-≤10 years of age) (Experimental): Subjects, who had previously received 1 injection of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine at 2-5 years of age, were administered 1 injection of the same vaccine at 7-10 years of age.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine
- Vaccine naive (≥7-≤10 years of age) (Experimental): Vaccine naive subjects, age-matched to the ≥7-≤10 years of age groups, received 1 injection of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine
- MenACWY-CRM_1 (≥11-≤15 years of age) (Experimental): Subjects, who had previously received 1 injection of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine at 7-10 years of age, were administered 1 injection of the same vaccine at 11-15 years of age.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine
- Vaccine naive (≥11-≤15 years of age) (Experimental): Vaccine naive subjects, age-matched to the ≥11-≤15 years of age group, received 1 injection of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine — Subjects received at day 1 a single dose of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine.

SUMMARY:
In this extension study, V59P20E1, the sponsor was planning to assess 5-year antibody persistence in subjects who received one or two doses of MenACWY conjugate vaccine at 2 to 10 years of age, and to evaluate response to a booster dose administered 5 years after primary vaccination in the parent study V59P20 (NCT00616421).

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, all subjects must meet ALL of the inclusion criteria described.

1. Subject has (a) parent(s) or legal guardian(s) who has/have given written consent after the nature of the study has been explained according to local regulatory requirements.
2. If the subject is of an age where, according to local regulations, informed assent is required, that subject has provided assent to participate in the study.
3. Subject is in good health as determined by the outcome of medical history, physical examination, and clinical judgment of the investigator.
4. A negative urine pregnancy test is required before female subjects of childbearing potential will be enrolled. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
5. For subjects who participated in study V59P20 (Groups MenACWYCRM_ 2 (≥7-≤10 Years), MenACWYCRM_1 (≥7-≤10 Years) and MenACWYCRM_ 1 (≥11-≤15 Years) only):

   * subject who enrolled in Groups MenACWYCRM_2 (≥7-≤10 Years), MenACWYCRM_1 (≥7-≤10 Years) and MenACWYCRM_1 (≥11-≤15 Years) of study V59P20, has completed this study and included in per protocol immunogenicity analysis;
   * the date of first vaccination in study V59P20 occurred 54 to 66 months prior to the collection of the blood sample at Visit 1.
6. For vaccine-naive subjects (Groups Vaccine Naive(≥7-≤10Years) and Vaccine Naive (≥11-≤15 Years) only):

   * Individual is a male or female 7 to 10 years of age (group Vaccine Naive(≥7-≤10Years)) or 11 to 15 years of age (Group Vaccine Naive (≥11-≤15 Years)).

Exclusion Criteria:

In order to participate in this study, all subjects must meet NONE of the exclusion criteria described.

1. If the subject is female of childbearing potential, sexually active, and has not used any of the acceptable contraceptive methods for at least 2 months prior to study entry and for the duration of the trial.
2. Subject is a pregnant or breast-feeding female.
3. Subjects' parents or legal guardians or subjects who are not able to comprehend and to follow all required study procedures for the whole period of the study.
4. History of documented or suspected invasive meningococcal disease.
5. Previous household contact with and/or intimate exposure to an individual with laboratory proven N. meningitidis infection within 60 days prior to enrollment and for the duration of the study.
6. Have received any other meningococcal vaccine since participation in V59P20 or, if vaccine-naive subjects, have not received any meningococcal vaccine since birth.
7. Suspected or known hypersensitivity reaction after a previous dose of Menveo, any component of this vaccine, including any other CRM197 and diphtheria toxoid.
8. Any contraindication or precaution against vaccination with Novartis Menveo™ vaccine as highlighted in the package insert.
9. Serious, chronic, or acute illnesses or diseases (i.e., cardiac, renal, neurologic, rheumatologic, metabolic, gastrointestinal, psychiatric, or other organ system).
10. Any confirmed or suspected condition with impaired/altered function of immune system (immunodeficient or autoimmune conditions).
11. Administration of any cancer chemotherapy, immune-modified or immunosuppressive agents or systemic corticosteroids for at least seven days at any dose in the past 12 weeks or planned use throughout the study period (nasal or inhaled steroids are permitted, as are steroids applied to the skin).
12. Administration of blood, blood products and/or plasma derivatives or any immunoglobulin preparation in the past 12 weeks or planned use throughout the study period.
13. Administration of any vaccine within 28 days prior to the study enrollment or planned administration during the study period.
14. Subjects participating in any clinical trial with another investigational product 28 days prior to first study visit or intent to participate in another clinical study at any time during the study period.
15. Subjects who have experienced a significant acute infection requiring systemic antibiotic treatment within the 5 days prior to enrolment or have experienced a body temperature ≥38°C (≥100.4°F) within the 3 days before the intended study vaccination.
16. Any condition which, in the opinion of the investigator, would pose a health risk to the participant.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 465 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (16):
- United States (15):
  - 82 Children s Inv Research Prgm (ChIRP) 2900 Medical Center Parkway, Ste. 300, Bentonville, Arkansas
  - 83 AR Pediatric Clinical Research 500 South University, Ste. 200, Little Rock, Arkansas
  - 32 Prem Health Research Center 9317 Firestone Blvd., Downey, California
  - 27 KY Pediatric Adult Research 201 South 5th Street, Suite 102, Bardstown, Kentucky
  - 36 Meridian Clinical Research 3319 N. 107th Street, Omaha, Nebraska
  - 33 Dr. Sender's and Associates 2054 South Green Road, Cleveland, Ohio
  - 31 Benchmark Research, Fort Worth 4504 Boat Club Rd., Suite 400A, Fort Worth, Texas
  - 25 Benchmark Research, San Angelo 3555 Knickerbocker Rd., San Angelo, Texas
  - 65 Westside Medical 1477 N 2000 W, Suite C, Clinton, Utah
  - 29 J. Lewis Research, Inc. 6360 South 3000 East, Ste. 100, Salt Lake City, Utah
  - 30 J. Lewis Research, Inc. 6360 South 3000 East, Ste. 100, Salt Lake City, Utah
  - 37 Copperview Medical Associates 3556 West 9800 South, South Jordan, Utah
  - 47 Wee Care Pediatrics 1792 W. 1700 S., Syracuse, Utah
  - 34 Rockwood Clinic P S 400 East Fifth Avenue, Spokane, Washington
  - 35 Rockwood Clinic-North Pediatrics 9001 N Country Homes Blvd, Spokane, Washington
- 26 Benchmark Research 3800 Houma Blvd., Suite 345, Metairie, LA, Ukraine

REFERENCES:
- [Background] Halperin SA, Gupta A, Jeanfreau R, Klein NP, Reisinger K, Walter E, Bedell L, Gill C, Dull PM. Comparison of the safety and immunogenicity of an investigational and a licensed quadrivalent meningococcal conjugate vaccine in children 2-10 years of age. Vaccine. 2010 Nov 23;28(50):7865-72. doi: 10.1016/j.vaccine.2010.09.092. Epub 2010 Oct 29. PMID 20943209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 22 study sites.
Pre-assignment Details: All subjects were included in the trial.
Groups:
- MenACWY-CRM_2 (≥7-≤10 Years): Subjects who had previously received 2 injections of MenACWY-CRM vaccine at 2-5 years of age, were administered 1 injection of MenACWY-CRM vaccine at 7-10 years of age.
- MenACWY-CRM_1 (≥7-≤10 Years): Subjects who had previously received 1 injection of MenACWY-CRM vaccine at 2-5 years of age, were administered 1 injection of MenACWY-CRM vaccine at 7-10 years of age.
- Vaccine Naive (≥7-≤10 Years): Vaccine naive subjects, age-matched to the ≥7-≤10 years of age groups, received 1 injection of MenACWY-CRM vaccine.
- MenACWY-CRM_1 (≥11-≤15 Years): Subjects who had previously received 1 injection of MenACWY-CRM vaccine at 6-10 years of age, were administered 1 injection of MenACWY-CRM vaccine at 11-15 years of age.
- Vaccine Naive (≥11-≤15 Years): Vaccine naive subjects, age-matched to the ≥11-≤15 years of age group, received 1 injection of MenACWY-CRM vaccine.
- Not Assigned: Two subjects 2-5 years of age were randomized to receive another meningococcal ACWY vaccine (not the investigational product in the extension study) in the parent study and therefore not eligible for enrolment into the extension study. These subjects were inadvertently enrolled and completed the extension study. During analysis, these two subjects were included in a separate "not assigned" group in the Full Analysis Set and excluded from the Per Protocol Set. However, one of these subjects actually received the investigational vaccine (due to a randomization error) in the parent study and was included in the safety analyses under MenACWY-CRM_1 (≥7-≤10 Years) group in the extension study.
Period: Overall Study
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | Vaccine Naive (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years) | Vaccine Naive (≥11-≤15 Years) | Not Assigned
Started | 73 | 103 | 120 | 66 | 101 | 2
Completed | 71 | 101 | 119 | 64 | 99 | 2
Not Completed | 2 | 2 | 1 | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Visit 1 delayed, unable to reschedule | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Met exclusion criterion No 6 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject moved out of the state | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was done on the all enrolled population.
Groups:
- Not Assigned: Two subjects 2-5 years of age were randomized to receive another meningococcal ACWY vaccine (not the investigational product in the extension study) in the parent study and therefore not eligible for enrolment into the extension study. These subjects were inadvertently enrolled and completed the extension study. During analysis, these two subjects were included in a separate "not assigned" group in the FAS and excluded from the PPS. However, one of these subjects actually received the investigational vaccine (due to a randomization error) in the parent study and was included in the safety analyses under MenACWY-CRM_1 (≥7-≤10 Years) group in the extension study.
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | Vaccine Naive (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years) | Vaccine Naive (≥11-≤15 Years) | Not Assigned | Total
Number analyzed (Participants) | 73 | 103 | 120 | 66 | 101 | 2 | 465
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (1.1) | 8.1 (1.2) | 8.5 (1.1) | 13.0 (1.6) | 11.8 (1.0) | 8.0 (1.4) | 9.7 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 49 | 63 | 28 | 46 | 1 | 222
  Male | 38 | 54 | 57 | 38 | 55 | 1 | 243

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Persisting hSBA Titers ≥1:8 Against Neisseria Meningitidis (N. Meningitidis) Serogroups A, C, W and Y, Five Years After Having Received One or Two Doses of MenACWY-CRM Vaccine
Description: The percentages of subjects with persisting serum bactericidal antibody ≥1: 8, against N.meningitidis serogroups A, C, W and Y, after having received one or two doses of MenACWY-CRM vaccine, five years earlier in the parent study, are reported.
  The serum bactericidal antibodies directed against N.meningitidis serogroups, are measured by human complement Serum Bactericidal Assay (hSBA).
Time Frame: 5 years post-vaccination
Population: The analysis was done on per-protocol population i.e all subjects who provided immunogenicity data; had no major protocol deviations and who were not excluded due to other reasons defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years)
Number analyzed (Participants) | 70 | 96 | 64
Percentages of subjects
  Serogroup A (N=68, 96, 64) | 7 [2 to 16] | 14 [7 to 22] | 22 [13 to 34]
  Serogroup C (N= 69, 96, 64) | 48 [36 to 60] | 32 [23 to 43] | 56 [43 to 69]
  Serogroup W (N= 69, 96, 64) | 83 [72 to 91] | 74 [64 to 82] | 80 [68 to 89]
  Serogroup Y | 50 [38 to 62] | 48 [38 to 58] | 53 [40 to 66]

2. Secondary Outcome: Persisting Geometric Mean Titers Against N.Meningitidis Serogroups A, C, W and Y in Subjects, Five Years After Having Received One or Two Doses of MenACWY-CRM Vaccine.
Description: The persistence of geometric mean titers (GMTs) against N.meningitidis serogroups A, C, W and Y in subjects who had received one or two doses of MenACWY-CRM vaccine, five years earlier in the parent study, are reported.
Time Frame: 5 years post-vaccination
Population: The analysis was done on per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years)
Number analyzed (Participants) | 70 | 96 | 64
Titers
  Serogroup A (N=68, 96, 64) | 2.41 [2.09 to 2.78] | 2.95 [2.42 to 3.61] | 3.73 [2.74 to 5.06]
  Serogroup C (N= 69, 96, 64) | 7.55 [5.44 to 10] | 6.5 [4.75 to 8.9] | 12 [7.72 to 19]
  Serogroup W (N= 69, 96, 64) | 23 [17 to 31] | 19 [14 to 25] | 26 [18 to 38]
  Serogroup Y | 8.57 [6.08 to 12] | 8.13 [6.11 to 11] | 10 [6.51 to 16]

3. Secondary Outcome: Percentages of Subjects With Persisting hSBA Titers ≥1:8 Against N.Meningitidis Serogroups A, C, W and Y as Compared to Age Matched Vaccine-naive Subjects
Description: The percentages of subjects with persisting serum bactericidal antibody ≥1: 8, against N.meningitidis serogroups A, C, W and Y, after having received one or two doses of MenACWY-CRM vaccine five years earlier in the parent study, are compared with the hSBA response in age matched vaccine-naive subjects.
Time Frame: 5 years post-vaccination; baseline for naive
Population: The analysis was done on per-protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | Vaccine Naive (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years) | Vaccine Naive (≥11-≤15 Years)
Number analyzed (Participants) | 70 | 96 | 118 | 64 | 100
Percentages of subjects
  Serogroup A (N= 68, 96, 118, 64, 100) | 7 [2 to 16] | 14 [7 to 22] | 0 [0 to 3] | 22 [13 to 34] | 5 [2 to 11]
  Serogroup C (N= 69, 96, 118, 64, 99) | 48 [36 to 60] | 32 [23 to 43] | 21 [14 to 30] | 56 [43 to 69] | 21 [14 to 31]
  Serogroup W (N= 69, 96, 118, 64, 100) | 83 [72 to 91] | 74 [64 to 82] | 52 [42 to 61] | 80 [68 to 89] | 54 [44 to 64]
  Serogroup Y | 50 [38 to 62] | 48 [38 to 58] | 23 [16 to 32] | 53 [40 to 66] | 37 [28 to 47]

4. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥1:8 Against N.Meningitidis Serogroups A, C, W and Y, After Receiving One Injection of MenACWY-CRM Vaccine in the Present Study.
Description: The antibody response against N.meningitidis serogroups A, C, W and Y, at one month after one injection of Men ACWY-CRM vaccine was administered in the present study to subjects who had received either one or two doses of MenACWY-CRM vaccine 5 years earlier and to age matched naive subjects, is evaluated in terms of the percentages of subjects with hSBA titers ≥1:8.
Time Frame: Day 28 post-vaccination
Population: The analysis was done on per-protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | Vaccine Naive (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years) | Vaccine Naive (≥11-≤15 Years)
Number analyzed (Participants) | 65 | 95 | 110 | 60 | 85
Percentages of subjects
  Serogroup A (N= 63, 95, 109, 60, 85) | 98 [91 to 100] | 100 [96 to 100] | 75 [66 to 83] | 100 [94 to 100] | 80 [70 to 88]
  Serogroup C (N= 65, 94, 109, 60, 85) | 100 [94 to 100] | 100 [96 to 100] | 82 [73 to 88] | 100 [94 to 100] | 86 [77 to 92]
  Serogroup W (N= 63, 95, 110, 60, 85) | 100 [94 to 100] | 100 [96 to 100] | 94 [87 to 97] | 100 [94 to 100] | 92 [84 to 97]
  Serogroup Y (N= 65, 94, 110, 59, 85) | 100 [94 to 100] | 100 [96 to 100] | 85 [77 to 91] | 100 [94 to 100] | 82 [73 to 90]

5. Secondary Outcome: Geometric Mean Titers Against N.Meningitidis Serogroups A, C, W and Y, After Receiving One Injection of MenACWY-CRM Vaccine in the Present Study.
Description: The antibody response against N.meningitidis serogroups A, C, W and Y, at one month after one injection of Men ACWY-CRM vaccine was administered in the present study to subjects who had received either one or two doses of MenACWY-CRM vaccine 5 years earlier and to age matched naive subjects, is evaluated in terms of GMTs.
Time Frame: Day 28 post-vaccination
Population: The analysis was done on per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | Vaccine Naive (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years) | Vaccine Naive (≥11-≤15 Years)
Number analyzed (Participants) | 65 | 95 | 110 | 60 | 85
Titers
  Serogroup A (N= 63, 95, 109, 60, 85) | 321 [241 to 428] | 361 [299 to 436] | 28 [20 to 39] | 350 [265 to 463] | 31 [22 to 45]
  Serogroup C (N= 65, 94, 109, 60, 85) | 760 [545 to 1059] | 498 [406 to 610] | 48 [33 to 70] | 712 [490 to 1036] | 102 [63 to 166]
  Serogroup W (N= 63, 95, 110, 60, 85) | 1571 [1247 to 1980] | 1534 [1255 to 1873] | 55 [42 to 72] | 1556 [1083 to 2237] | 69 [48 to 99]
  Serogroup Y (N= 65, 94, 110, 59, 85) | 1286 [992 to 1668] | 1693 [1360 to 2107] | 48 [34 to 66] | 1442 [1050 to 1979] | 45 [30 to 69]

6. Secondary Outcome: Number of Subjects Reporting Solicited Adverse Events, After Receiving One Injection of MenACWY-CRM Vaccine in the Present Study.
Description: The number of subjects reporting solicited local and systemic adverse events after one injection of MenACWY-CRM vaccine was administered in the present study to,
  1. Subjects, who had 5 years earlier received either one or two doses of MenACWY-CRM vaccine
  2. Vaccine-naive subjects.
Time Frame: Day 1 to day 7 post-vaccination
Population: The analysis was done on solicited safety set, ie, all subjects in the exposed set who provided post vaccination solicited reactogenicity data.
Measure: Number; unit: Number of subjects
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | Vaccine Naive (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years) | Vaccine Naive (≥11-≤15 Years)
Number analyzed (Participants) | 69 | 100 | 119 | 64 | 98
Number of subjects
  Injection site pain (N= 68, 99, 117, 64, 98) | 39 | 52 | 42 | 31 | 47
  Injection site erythema (N= 68, 99, 117, 64, 98) | 10 | 13 | 10 | 10 | 6
  Injection site induration (N= 68, 99, 119, 64, 98) | 12 | 12 | 7 | 7 | 8
  Chills (N= 68, 99, 117, 64, 98) | 5 | 3 | 6 | 1 | 2
  Malaise (N= 69, 99, 117, 64, 98) | 15 | 14 | 13 | 11 | 19
  Myalgia (N= 69, 99, 117, 64, 98) | 9 | 8 | 8 | 4 | 8
  Arthralgia (N= 69, 99, 117, 64, 98) | 8 | 4 | 5 | 4 | 8
  Headache (N= 69, 99, 117, 64, 97) | 13 | 9 | 22 | 12 | 21
  Nausea (N= 68, 99, 117, 64, 97) | 10 | 11 | 12 | 7 | 8
  Fever (≥38°C; N= 66, 99, 115, 64, 96) | 1 | 0 | 3 | 1 | 0
  Prophyl. use analg/antip (N= 68, 99, 118, 63, 97) | 0 | 1 | 2 | 1 | 1
  Thera. use anal/antipyret (N= 69, 99, 118, 64, 97) | 14 | 12 | 11 | 11 | 6

7. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events, After Receiving One Injection of MenACWY-CRM Vaccine in the Present Study.
Description: The safety and tolerability of one injection of MenACWY-CRM vaccine, administered in the present study, was evaluated in terms of the number of subjects reporting unsolicited adverse events, serious adverse events and adverse events leading to premature withdrawal.
Time Frame: Day 1 to day 28
Population: The analysis was done on unsolicited safety set, ie, all exposed subjects who provided unsolicited adverse events (AE) data.
Measure: Number; unit: Number of subjects
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | Vaccine Naive (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years) | Vaccine Naive (≥11-≤15 Years)
Number analyzed (Participants) | 73 | 102 | 120 | 65 | 100
Number of subjects
  Any adverse event (AE) | 18 | 23 | 19 | 18 | 11
  Possibly/Probably related unsolicited AE | 4 | 3 | 4 | 7 | 5
  Any SAE | 0 | 0 | 1 | 0 | 1
  Possibly/Probably related SAE | 0 | 0 | 0 | 0 | 0
  AE leading to withdrawal | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All solicited AE were collected from day 1 to day 7; unsolicited AEs, AE's leading to premature withdrawal and all Serious Adverse Events were collected throughout the study (day1 to day 28).
Description: All solicited AEs are reported as systematic assessment ; all unsolicited AEs are reported as non-systematic assessment.
  Serious adverse events analysis was done on the unsolicited safety set, other adverse events analysis was done on the overall safety set.
Arm/Group | MenACWY-CRM_2 (≥7-≤10 Years) | MenACWY-CRM_1 (≥7-≤10 Years) | Vaccine Naive (≥7-≤10 Years) | MenACWY-CRM_1 (≥11-≤15 Years) | Vaccine Naive (≥11-≤15 Years)
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/102 | 1/120 | 0/65 | 1/100
Other Adverse Events (participants affected / at risk) | 48/73 | 70/102 | 77/120 | 46/65 | 66/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM_2 (≥7-≤10 Years) (N=73) | MenACWY-CRM_1 (≥7-≤10 Years) (N=102) | Vaccine Naive (≥7-≤10 Years) (N=120) | MenACWY-CRM_1 (≥11-≤15 Years) (N=65) | Vaccine Naive (≥11-≤15 Years) (N=100)
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM_2 (≥7-≤10 Years) (N=73) | MenACWY-CRM_1 (≥7-≤10 Years) (N=102) | Vaccine Naive (≥7-≤10 Years) (N=120) | MenACWY-CRM_1 (≥11-≤15 Years) (N=65) | Vaccine Naive (≥11-≤15 Years) (N=100)
Nausea (Gastrointestinal disorders) | 12 | 12 | 14 | 8 | 9
Chills (General disorders) | 5 | 3 | 6 | 2 | 2
Injection site erythema (General disorders) | 25 | 34 | 28 | 17 | 21
Injection site induration (General disorders) | 21 | 26 | 26 | 17 | 17
Injection site pain (General disorders) | 42 | 57 | 51 | 34 | 52
Malaise (General disorders) | 15 | 14 | 13 | 12 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 5 | 5 | 4 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 13 | 10 | 4 | 9
Headache (Nervous system disorders) | 14 | 11 | 23 | 15 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.